CLINICAL TRIAL: NCT04867967
Title: Yoga and Mindfulnes-based-stress-reduction for Patients With Tension-type Headache
Brief Title: Yoga and MBSR for TTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Eden Stiftung (Unknown)
Responsible Party: Principal Investigator, Holger Cramer, PD Dr. rer. medic, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-7925 BO
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Tension-Type Headache
Keywords: Tension-Type Headache; Yoga; Mindfulness-based stress reduction
MeSH Terms: conditions — Tension-Type Headache | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iyengar Yoga Intervention (Experimental): 8-week yoga class; once weekly; 90 minutes
  Note: First administered face-to-face, due to Covid-restrictions changed to online classes
  Interventions: Behavioral: Iyengar Yoga
- Mindfulness-based stress reduction (Active Comparator): 8-week MBSR class; once weekly; 90 minutes
  Note: First administered face-to-face, due to Covid-restrictions changed to online classes
  Interventions: Behavioral: Mindfulness-based stress reduction
- Waitlist control (No Intervention): Waitlist control, ususal care

INTERVENTIONS:
Behavioral: Iyengar Yoga — Classical Iyengar Yoga intervention, especially designed for headache patients. Note: First administered face-to-face, due to Covid-restrictions changed to online classes
  Arms: Iyengar Yoga Intervention
Behavioral: Mindfulness-based stress reduction — Standardazied Mindfulness-based stress reduction intervention Note: First administered face-to-face, due to Covid-restrictions changed to online classes
  Arms: Mindfulness-based stress reduction

SUMMARY:
Primary study objectives

1. evaluate the short-term effect of yoga intervention in addition to routine care on headache frequency in patients with frequent or chronic tension-type headache compared to routine care alone (waiting group).
2. to evaluate the short-term effect of yoga intervention in addition to routine care on headache frequency in patients with frequent episodic or chronic tension-type headache compared with stress management through mindfulness-based stress reduction (MBSR) in addition to routine care.

Secondary study objectives

Evaluation of the medium-term effect of the intervention on headache frequency as well as the short- and medium-term effect on the secondary target parameters in comparison to the waiting group and MBSR. Further evaluation of the safety and acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* episodic or chronic tension-type headache according to ICHD-3 definition

Exclusion Criteria:

* medication induced headache according to ICHD-3 definition
* Cluster-headache according to ICHD-3 definition
* serious chronic systemic or acute physical or mental illness
* Dementia
* Pregnancy
* actual in a yoga or MBSR class

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Headache Frequency | post-intervention (8 weeks)
  Headache Frequency self-reported by a headache diary

SECONDARY OUTCOMES:
Headache Frequency | follow-up (20 weeks)
  Headache Frequency self-reported by a headache diary
Duration of headache episodes | post-intervention (8 weeks)
  Duration of headache episodes self-reported by a headache diary
Duration of headache episodes | follow-up (20 weeks)
  Duration of headache episodes self-reported by a headache diary
Pain Intensity | post-intervention (8 weeks)
  Numeric rating scale
Pain Intensity | follow-up (20 weeks)
  Numeric rating scale (NRS)
Pain medication use | post-intervention (8 weeks)
  Pain medication use self-reported by a headache diary
Pain medication use | follow-up (20 weeks)
  Pain medication use self-reported by a headache diary
Headache related disability | post-intervention (8 weeks)
  Headche Impact Test 6 (HIT-6)
Headache related disability | follow-up (20 weeks)
  Headche Impact Test 6 (HIT-6)
Health-related quality of life | post-intervention (8 weeks)
  SF-36 questionaire
Health-related quality of life | follow-up (20 weeks)
  SF-36 questionaire
Anxiety | post-intervention (8 weeks)
  Depression and Anxiety scale (DAAS)
Anxiety | follow-up (20 weeks)
  Depression and Anxiety scale (DAAS)
Stress | post-intervention (8 weeks)
  Depression and Anxiety scale (DAAS)
Stress | follow-up (20 weeks)
  Depression and Anxiety scale (DAAS)
Pain catastrophizing | post-intervention (8 weeks)
  Pain catastrophizing scale (PCS)
Pain catastrophizing | follow-up (20 weeks)
  Pain catastrophizing scale (PCS)
Pain acceptance | post-intervention (8 weeks)
  Chronic pain acceptance questionaire (CPAQ)
Pain acceptance | follow-up (20 weeks)
  Chronic pain acceptance questionaire (CPAQ)
Mindfulness | post-intervention (8 weeks)
  Mindfulness Attention and Awerness scale (MAAS)
Mindfulness | follow-up (20 weeks)
  Mindfulness Attention and Awerness scale (MAAS)
Body Awareness | post-intervention (8 weeks)
  Body Awareness questionaire (BAQ)
Body Awareness | follow-up (20 weeks)
  Body Awareness questionaire (BAQ)
Safety | post-intervention (8 weeks)
  Adverse events
Safety | follow-up (20 weeks)
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, MD, Study Chair — University of Duisburg-Essen, Faculty of Medicine
Locations (1):
- Evang. Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No